CLINICAL TRIAL: NCT06993987
Title: Study of Interactions Between Oncologists and Resuscitators to Optimize Decision Making for Admission of Patients With Metastatic Solid Cancer to the ICU
Brief Title: Study of Interactions Between Oncologists and Resuscitators to Optimize Decision Making for Admission of Patients With Metastatic Solid Cancer to the ICU (InterOncoRea)
Acronym: InterOncoRea
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC25.0045 - InterOncoRea
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-03

CONDITIONS: Intensive Care Unit (ICU) Patients; Metastatic Cancer
Keywords: Metastatic cancer; Intensive care; Admission of a patient with metastatic solid cancer to intensive care; Metastatic solid cancer and intensive care; Communication between intensivists and oncologists; Reason for hospitalization for patients with metastatic solid cancer; Survival for patients with metastatic cancer after admission to the intensive care unit; Metastatic solid cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with metastatic solid cancer admitted to the ICU
  Interventions: Other: Descriptive analysis

INTERVENTIONS:
Other: Descriptive analysis — The descriptive analysis of qualitative variables (reason for admission) will be carried out in the form of frequencies and percentages. Quantitative variables will be described in terms of averages, medians or standard deviations, as required.

SUMMARY:
The aim of our study is to optimise the interaction between oncologists and resuscitators to improve decision-making regarding the admission of patients with metastatic solid cancers to the ICU.

The study is structured into two successive stages. The first stage involves a retrospective descriptive analysis of patients with metastatic solid cancer admitted to the ICU, to enable comparison with centres that have already documented this subject.

The second stage involves personalised interviews with medical staff working in both the oncology department and the intensive care unit.

DETAILED DESCRIPTION:
In the vast majority of cases, there is no cure for metastatic solid cancer. As a result, the question of end of life is very often present.

End of life may be linked to the aggressiveness of the disease, to therapeutic damage, but also to an independent acute event that may occur during the course of oncology care.

This explains why the question of resuscitation management comes into play in the care of our oncology patients.

The literature shows that one in 7 patients admitted to intensive care in Europe has a history of cancer, and that 5 to 10% of cancer patients will require intensive care during their course of treatment.

The therapeutic advances brought about by immunotherapy in the first instance, followed by targeted therapies in a second phase, have considerably altered the prognosis of patients with solid cancers, including the most aggressive cancers.

However, given the poor prognosis of these diseases, having metastatic cancer continues to hinder a patient's possible admission to the intensive care unit.

The second most common reason for refusing admission to the ICU is having cancer.

Yet the post-ICU mortality rate for cancer patients is identical to that of the entire ICU patient group.

Various scores have been used to determine the 'right' criteria for ICU admission for patients with metastatic solid cancers.

Nevertheless, nothing appears to be more effective than communication between oncologists and intensive care physicians, particularly since the prognosis of patients with advanced cancers is still a subject of interdisciplinary discussion.

Various scores have attempted to establish the 'right' criteria for admitting patients with metastatic solid cancers to intensive care.

However, nothing appears more effective than discussions between oncologists and resuscitators, particularly given that the prognosis of patients with advanced cancers is still a topic of interdisciplinary debate.

Indeed, the decision to admit a patient with metastatic cancer to an intensive care unit appears to raise ethical, medical and organisational issues.

Bearing this in mind, and given the numerous studies already conducted in this area, we thought it would be interesting to examine the relationship between oncology and intensive care units.

To study the interactions between intensive care physicians and oncologists and identify areas for improvement in patient care, we devised a two-stage approach.

First, we conducted personalised semi-structured interviews with doctors from the medical oncology department (oncologists, organ specialists and general practitioners) and doctors from the intensive care unit. This allowed us to identify the obstacles that each speciality faces when admitting a patient to the intensive care unit. This would enable us to deduce the elements essential for reaching an agreement on admitting a patient to the intensive care unit (Stage 1).

Secondly, we will review practices at Brest University Hospital (and possibly other centres that might be interested in our work) and compare them with data in the literature to see if our decisions are similar to those made in other centres that have already documented the subject (Stage 2).

ELIGIBILITY:
Inclusion Criteria:

* Major patient hospitalized in medical or surgical intensive care with metastatic solid cancer, whatever the primary site and whatever the reason for admission to the intensive care unit
* Start of stay in intensive care must be between June 1, 2023 and June 1, 2024.

Exclusion Criteria:

* Patient objecting to data processing
* The patient is under legal protection (e.g. guardianship or curatorship)
* A patient with multiple synchronous cancers
* Diagnosis of metastatic cancer during stay in intensive care unit intensive care unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients with metastatic solid cancer
Sampling Method: Non-Probability Sample
Enrollment: 139 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of reason for admission to intensive care unit | Patients admitted to intensive care between June 1, 2023 and June 1, 2024.
  Analysis of the reason for admission to intensive care unit

SECONDARY OUTCOMES:
Protective and risk factors | Patients admitted to intensive care between June 1, 2023 and June 1, 2024.
  Protective and risk factors for returning home within 3 months
Survival at 1 month and 3 months | Patients admitted to intensive care between June 1, 2023 and June 1, 2024.
  Survival at 1 month and 3 months from admission to intensive care unit
Risk factors for survival in intensive care | Patients admitted to intensive care between June 1, 2023 and June 1, 2024.

OTHER OUTCOMES:
Criteria for ICU admission of patients | Patients admitted to intensive care between June 1, 2023 and June 1, 2024.
  Identification and categorization of major decision criteria reported by physicians for ICU admission of patients with metastatic solid cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement

REFERENCES:
- [Result] Iapichino G, Corbella D, Minelli C, Mills GH, Artigas A, Edbooke DL, Pezzi A, Kesecioglu J, Patroniti N, Baras M, Sprung CL. Reasons for refusal of admission to intensive care and impact on mortality. Intensive Care Med. 2010 Oct;36(10):1772-1779. doi: 10.1007/s00134-010-1933-2. Epub 2010 Jun 9. PMID 20533023
- [Result] Robert R, Reignier J, Tournoux-Facon C, Boulain T, Lesieur O, Gissot V, Souday V, Hamrouni M, Chapon C, Gouello JP; Association des Reanimateurs du Centre Ouest Group. Refusal of intensive care unit admission due to a full unit: impact on mortality. Am J Respir Crit Care Med. 2012 May 15;185(10):1081-7. doi: 10.1164/rccm.201104-0729OC. Epub 2012 Feb 16. PMID 22345582
- [Result] Padhi S, Shrestha P, Alamgeer M, Stevanovic A, Karikios D, Rajamani A, Subramaniam A. Oncology and intensive care doctors' perception of intensive care admission of cancer patients: A cross-sectional national survey. Aust Crit Care. 2024 Jul;37(4):520-529. doi: 10.1016/j.aucc.2023.12.005. Epub 2024 Feb 12. PMID 38350752
- [Result] Nassar AP Jr, Dettino ALA, Amendola CP, Dos Santos RA, Forte DN, Caruso P. Oncologists' and Intensivists' Attitudes Toward the Care of Critically Ill Patients with Cancer. J Intensive Care Med. 2019 Oct;34(10):811-817. doi: 10.1177/0885066617716105. Epub 2017 Jul 5. PMID 28675982
- [Result] Toffart AC, Gonzalez F, Hamidfar-Roy R, Darrason M. [ICU admission for cancer patients with respiratory failure: An ethical dilemma]. Rev Mal Respir. 2023 Oct;40(8):692-699. doi: 10.1016/j.rmr.2023.07.003. Epub 2023 Aug 31. French. PMID 37659881
- [Result] Borcoman E, Dupont A, Mariotte E, Doucet L, Joseph A, Chermak A, Valade S, Resche-Rigon M, Azoulay E, Lemiale V. One-year survival in patients with solid tumours discharged alive from the intensive care unit after unplanned admission: A retrospective study. J Crit Care. 2020 Jun;57:36-41. doi: 10.1016/j.jcrc.2020.01.027. Epub 2020 Jan 30. PMID 32032902
- [Result] Gwilliam B, Keeley V, Todd C, Roberts C, Gittins M, Kelly L, Barclay S, Stone P. Prognosticating in patients with advanced cancer--observational study comparing the accuracy of clinicians' and patients' estimates of survival. Ann Oncol. 2013 Feb;24(2):482-488. doi: 10.1093/annonc/mds341. Epub 2012 Oct 1. PMID 23028038
- [Result] Miller KD, Nogueira L, Devasia T, Mariotto AB, Yabroff KR, Jemal A, Kramer J, Siegel RL. Cancer treatment and survivorship statistics, 2022. CA Cancer J Clin. 2022 Sep;72(5):409-436. doi: 10.3322/caac.21731. Epub 2022 Jun 23. PMID 35736631
- [Result] Bos MM, Verburg IW, Dumaij I, Stouthard J, Nortier JW, Richel D, van der Zwan EP, de Keizer NF, de Jonge E. Intensive care admission of cancer patients: a comparative analysis. Cancer Med. 2015 Jul;4(7):966-76. doi: 10.1002/cam4.430. Epub 2015 Apr 18. PMID 25891471
- [Result] Puxty K, McLoone P, Quasim T, Sloan B, Kinsella J, Morrison DS. Risk of Critical Illness Among Patients With Solid Cancers: A Population-Based Observational Study. JAMA Oncol. 2015 Nov;1(8):1078-85. doi: 10.1001/jamaoncol.2015.2855. PMID 26313462
- [Result] Taccone FS, Artigas AA, Sprung CL, Moreno R, Sakr Y, Vincent JL. Characteristics and outcomes of cancer patients in European ICUs. Crit Care. 2009;13(1):R15. doi: 10.1186/cc7713. Epub 2009 Feb 6. PMID 19200368